CLINICAL TRIAL: NCT05376683
Title: Personalised Continuous Dose Titration of Combination Therapy for Hypertension Using CURATE: AI Personalised Continuous Dose Titration Platform
Brief Title: AI for Anti-hypertensive Medication Titration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandra Hospital (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Laureen Yi-Ting Wang, Principal investigator, Alexandra Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2022/00115
Record Dates: First submitted 2022-04-23; First posted 2022-05-17 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a 3 armed study.
  1. Control = SOC, 15 participants
  2. CURATE.AI (device)+telemonitoring= 15 participants.
  3. Telemonitoring without CURATE.AI= 15 participants. The rationale for the 3rd arm is that the process of telemonitoring itself can result in behavior change and affect blood pressure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Telemonitoring group (Active Comparator)
  Interventions: Behavioral: Telemonitoring
- AI. + Telemonitoring group (Active Comparator)
  Interventions: Device: Curate.AI; Behavioral: Telemonitoring

INTERVENTIONS:
Device: Curate.AI — Personalized, continuous recommendations on anti-hypertensive medication dose titration using an AI-derived platform also known as Curate.AI
  Arms: AI. + Telemonitoring group
Behavioral: Telemonitoring — Patients will report their blood pressure to a telemonitoring health platform
  Arms: AI. + Telemonitoring group; Telemonitoring group

SUMMARY:
Hypertension - a chronic condition of elevated blood pressure (BP) - is a highly prevalent condition. However, effective prevention and management of hypertension remain challenging under the current standard of care (SOC). There has been a growing recognition that one-off, irregular office BP measurements are not sufficient and that regular home BP monitoring will likely be an adjunct to conventional office BP measurements. By using artificial intelligence (AI), via the CURATE.AI platform, the goal is to use patients' BP data to rapidly generate personalized anti-hypertensive dose titrations. The main aim of this study is to assess the feasibility of CURATE.AI-assisted dose titration.

DETAILED DESCRIPTION:
The primary aim is to assess the feasibility of CURATE.AI-assisted dose titration intervention (daily home BP monitoring via telemonitoring BotMD Care platform combined with personalized continuous dose titration based on CURATE.AI recommendations to treating physicians).

The secondary objective is to evaluate the safety and generate estimates of effect size using a small three-arm study design (N=45; 1:1:1 randomization), to inform the power analysis and sample size calculation for a larger randomized controlled trial (RCT) evaluating the efficacy and safety of the CURATE.AI-assisted dose titration intervention. The other aim is to also understand the potential efficacy of the CURATE.AI-assisted dose titration intervention to improve treatment efficacy outcomes.

The investigators hypothesize that it will be logistically and scientifically feasible to use CURATE.AI-assisted dose titration for the management of hypertension,

ELIGIBILITY:
Inclusion Criteria:

* At least >=30 years of age and <=80 years
* History of uncontrolled primary hypertension, BPs more >=140/90mm Hg, treatment-naive or on single antihypertensive medication
* Not known to have complications of hypertension
* Sufficiently fluent in English language
* Able to give informed consent
* eGFR > 60 ml/min
* Eligible to undergo CCB + ARB/ACE-i therapy for =30 days

Exclusion Criteria:

* Suspected or known secondary hypertension
* Drug allergies to anti-hypertensive agents or agents of the same drug class used in the protocol
* Known postural hypotension or standing systolic blood pressure < 110 mmHg
* Malignant hypertension (BPs = 180/110 mmHg) that requires emergency treatment
* Arm circumference that does not fit BP cuff size which can affect the accuracy of BP measurement
* Pregnant women, trying to become pregnant or of child-bearing potential and not using birth control
* History of cancer
* Chronic kidney disease (eGFR <50ml/min) or end stage renal failure
* Liver cirrhosis or hepatic failure
* Chronic heart failure
* Chronic lung disease
* Diabetes Mellitus on insulin and/or with microvascular/macrovascular complications.
* Established cardiovascular disease such as stroke/transient ischemic attack and ischemic heart disease
* Potential psychosocial factors or serious medical conditions limiting the ability to self-monitor their blood pressure or limit adherence to interventions (E.g. dementia, active substance abuse, nursing home resident)
* Participants without informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Logistical feasibility of a protocol using telemonitoring and CURATE.AI-assisted dose titration. | 30 days
  A composite of the percentages will be use to obtain overall logistical feasibility of the protocol
  * BP monitoring adherence: Percentage of BP entries by participants into telehealth platform
  * Drug dose adherence percentage
  * Physician acceptability of CURATE.AI dose recommendations: the percentage of CURATE.AI recommended doses that were prescribed by the treating physician(s)
Scientific Feasibility | 30 days
  A composite of the percentages will be use to obtain overall scientificl feasibility of the protocol
  * CURATE.AI applicability: percentage of participants in whom CURATE.AI profiles can be generated and applied
  * Percentage of dosing cycles, out of 10 dosing cycles, that CURATE.AI recommends dose with calibration and efficacy intent to physicians
  * Percentage of participants with clinically significant dose changes: the cumulative dose is substantially (≥10%) different from the projected standard of care cumulative dose

SECONDARY OUTCOMES:
Generate pilot efficacy of telemonitoring and CURATE.AI-assisted dose titration protocol. | 3 months
  Mean change and time taken for in office BP between baseline and 1-month clinic visit towards reaching the target office systolic BP<140mmHg and diastolic BP<90mmHg.
Generate pilot efficacy of telemonitoring and CURATE.AI-assisted dose titration protocol. | 3 months
  -Percentage of participants with office systolic BP<140mmHg and/OR diastolic BP<90mmHg at 1-month.
Generate pilot efficacy of telemonitoring and CURATE.AI-assisted dose titration protocol. | 3 months
  -Time in therapeutic range: the percentage of home BP measurements recorded within the target home range during the CURATE.AI-assisted efficacy-driven dose recommendation stage
Generate pilot safety data of telemonitoring and CURATE.AI-assisted dose titration protocol. | 3 months
  The composite of hospitalizations due to hypotension, bradycardia, hyperkalemia, or acute kidney injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blasiak A, Khong J, Kee T. CURATE.AI: Optimizing Personalized Medicine with Artificial Intelligence. SLAS Technol. 2020 Apr;25(2):95-105. doi: 10.1177/2472630319890316. Epub 2019 Nov 26. PMID 31771394
- [Derived] Truong ATL, Tan SB, Wang GZ, Yip AWJ, Egermark M, Yeung W, Lee VV, Chan MY, Kumar KS, Tan LWJ, Vijayakumar S, Blasiak A, Wang LYT, Ho D. CURATE.AI-assisted dose titration for anti-hypertensive personalized therapy: study protocol for a multi-arm, randomized, pilot feasibility trial using CURATE.AI (CURATE.AI ADAPT trial). Eur Heart J Digit Health. 2023 Oct 24;5(1):41-49. doi: 10.1093/ehjdh/ztad063. eCollection 2024 Jan. PMID 38264697